CLINICAL TRIAL: NCT06509464
Title: Response Of Metabolic Syndrome Severity Score To High Intenisty Interval Training In Women With Central Obesity.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Soma Adel Gaber Abd El-Ghany (Other)
Responsible Party: Sponsor-Investigator, Soma Adel Gaber Abd El-Ghany, Assistant Lecturer, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cairo soma 46
Record Dates: First submitted 2024-07-09; First posted 2024-07-19 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Metabolic Syndrom
Keywords: Metabolic syndrom severity score; Metabolic syndrom; Central obesity
MeSH Terms: conditions — Obesity, Abdominal | interventions — Caloric Restriction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low volume High-intensity interval training (HIIT) (Experimental): group A (n =24) will receive low volume High-intensity interval training (HIIT) three times /week for 3 months,
  Interventions: Device: High intensity interval training; Dietary Supplement: Caloric restricted diet
- caloric restricted diet. (Experimental): group B (24) will receive caloric restricted diet.
  Interventions: Device: High intensity interval training; Dietary Supplement: Caloric restricted diet

INTERVENTIONS:
Device: High intensity interval training — High intensity interval training on treadmill
Dietary Supplement: Caloric restricted diet — Caloric restricted diet

SUMMARY:
This study will be conducted to investigate any significant effect of high intensity interval training on metabolic syndrome severity score in women with central obesity.

DETAILED DESCRIPTION:
RESPONSE OF METABOLIC SYNDROME SEVERITY SCORE TO HIGH INTENISTY INTERVAL TRAINING IN WOMEN WITH CENTRAL OBESITY

forty eight women with age ranges from 25 to 45 years old will be selected from nutrition-outpatient clinic; they will participate in the study for 6 weeks, and randomly be assigned into two equal groups.

Study group A (n =24) will receive low volume High-intensity interval training (HIIT) three times /week for 6 weeks , study group B (n =24) will receive caloric restriction diet

For evaluation Physical efficiency index using Modified Harvard Step test It is a powerful indicator for aerobic fitness. The Fitness Index score is determined according to the following equation

Fitness Index (long form) = (100 x test duration in seconds) divided by (2 x sum of heart beats in the recovery periods).

Metabolic syndrome severity score Metabolic syndrome severity score will be calculated through MetS Calculator (MetSCalc).

-3Laboratory investigation before & after treatment: for fasting blood glucose level and Lipid profile (total cholesterol, LDL, HDL, TAGs).

4- The 45-item Diet Satisfaction Questionnaire (DSat-45)

B) For treatment

1- Grand II Treadmill: (AC999- for maximum weight 150 Kg-

ELIGIBILITY:
Inclusion Criteria:

- 1. 48 Women subjects with age ranges from 25to 45 years.

2. Waist height ratio ranges from 49-58 (overweight and seriously overweight).

Exclusion Criteria:

* 1. Uncontrolled Diabetes 2. Uncontrolled hypertension 3. Cognitive impaired patients 4. Severe Anemic women 5. Subjects with physical or musculoskeletal disabilities 6. Pregnancy 7. Recent cardiothoracic surgery

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Metabolic syndrome severity score | 6weeks
Physical efficiency index using Modified Harvard Step test | 6weeks
The 45-item Diet Satisfaction Questionnaire (DSat-45 | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nesreen Ghareeb Elnahas, Professor, Principal Investigator — Cairo University
Locations (1):
- Faculty of physical therapy cairo university, Giza, Egypt